CLINICAL TRIAL: NCT03874923
Title: Comparison of 250 ml Versus 500 ml of Fluid Challenge on Oxygen Consumption in Critical Care Patients: an Open Label Multicentre Prospective Study
Brief Title: Comparison of 250 ml Versus 500 ml of Fluid Challenge
Acronym: KOBIAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0034
Record Dates: First submitted 2019-03-07; First posted 2019-03-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Fluid Challenge; Oxygen Consumption; Critical Care
Keywords: fluid expansion; oxygen delivery; tissue perfusion; cardiac output

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 250 mL of fluid challenge (Active Comparator)
  Interventions: Other: Fluid challenge
- 500 mL of fluid challenge (Experimental)
  Interventions: Other: Fluid challenge

INTERVENTIONS:
Other: Fluid challenge — After randomisation, patient will receive 250 ml or 500 ml of fluid challenge. VO2 will be assessed before fluid challenge, immediately, 30 minutes and 60 minutes after fluid challenge.

SUMMARY:
The objective of fluid challenge is to increase oxygen delivery (DO2) in order to improve/restore tissue oxygen consumption (VO2). However the fluid challenge volume to administer stills in debate, some studies recommend to administer 250 mL. Previous studies suggested that 500 mL of fluid challenge administration may improve cardiac output and oxygen delivery. The relation between the amount of fluid expansion and oxygen delivery and oxygen consumption was not yet been studied in a randomized study in critical care patients. This is the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient for whom the physician in charge decided to infuse fluid challenge because of signs of acute circulatory failure (systolic arterial blood pressure < 90mmHg, and/or mean arterial blood pressure< 65 mmHg, and/or the need of vasopressive amine infusion, and/or skin mottling, and/or diuresis <0.5 mL/kg/h for more than 2 hours, and/or arterial lactate level>2mmol/L.
* Echogenic patient
* Patient with a Stroke Volume (SV) variation with passive leg raising (PLR) more than 10%.
* Patient with regular sinus rhythm.
* Patient who received protocol information.

Exclusion Criteria:

* Age Under 18-year-old.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
VO2 after fluid challenge | 30 minutes after fluid challenge.
  Tissue oxygen consumption (VO2) after fluid challenge
VO2 after fluid challenge | 60 minutes after fluid challenge.
  Tissue oxygen consumption (VO2) after fluid challenge

SECONDARY OUTCOMES:
Change of arterial lactate concentration from baseline | 30 minutes after fluid challenge.
  Baseline is the measurement of arterial lactate concentration immediately after fluid challenge
Change of arterial lactate concentration from baseline | 60 minutes after fluid challenge.
  Baseline is the measurement of arterial lactate concentration immediately after fluid challenge
Respiratory variation of stroke volume | Immediately, 30 and 60 minutes after fluid challenge.
  Respiratory variation of stroke volume after fluid challenge.
PaO2/FiO2 | Immediately, 30 and 60 minutes after fluid challenge.
  PaO2/FiO2 ratio (ratio of arterial oxygen partial pressure to fractional inspired oxygen) after fluid challenge
Respiratory variation of the pulse pressure | 30 and 60 minutes after fluid challenge.
  Respiratory variation of the pulse pressure
Stroke volume variation with passive leg raising (PLV) | 30 and 60 minutes after fluid challenge.
  Stroke volume variation with passive leg raising (PLV)
Systolic heart function (LVEF) | Immediately, 30 and 60 minutes after fluid challenge.
  Systolic heart function (LVEF)
Diastolic heart function | Immediately, 30 and 60 minutes after fluid challenge.
  Diastolic heart function (E, A, E', A', S' waves)

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abou-Arab, Dr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No